CLINICAL TRIAL: NCT07111481
Title: Effect of Music on Surgical Performance During Artificial Intelligence Based Simulation Training: A Randomized Controlled Trial
Brief Title: Effect of Music on Surgical Performance During Artificial Intelligence-Based Simulation Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Rolando Del Maestro, Director, Neurosurgical Simulation and Artificial Intelligence Learning Centre, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2010-270, NEU-09-042-Trial 6
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-08

CONDITIONS: Surgical Education
Keywords: Neurosurgery; Virtual Reality; Surgical Simulation; Music; Mozart Effect; Artificial Intelligence; Intelligent Tutoring Systems

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: Study participants are blinded to group assignments and study outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No music group (No Intervention): 20 participants allocated. Participants perform a simulated subpial brain tumor resection on the NeuroVR simulator without music while receiving verbal feedback from the ICEMS tutor.
- Mozart music group (Experimental): 20 participants allocated. Participants will listen to Mozart music while performing a simulated subpial brain tumor resection on the NeuroVR simulator and receiving verbal feedback from the ICEMS tutor.
  Interventions: Behavioral: Mozart music

INTERVENTIONS:
Behavioral: Mozart music — Participants will be played Mozart's Sonata for Two Pianos in D Major, K. 448 during their surgical simulation training session with an AI tutor.
  Arms: Mozart music group

SUMMARY:
At the Neurosurgical Simulation and Artificial Intelligence Learning Centre, we seek to provide surgical trainees with innovative technologies that allow them to improve their surgical technical skills in risk-free environments, potentially improving patient operative outcomes. The Intelligent Continuous Expertise Monitoring System (ICEMS), a deep learning application that assesses and trains neurosurgical technical skill and provides continuous intraoperative feedback, is one such technology that may improve surgical education.

Previous research has found that music can impact cognitive performance and learning outcomes. However, the effects of music on neurosurgical simulation performance-along with the associated affective-cognitive responses-remain largely unexplored.

In this randomized controlled trial, medical students from four Quebec universities will be blinded and randomized to one of two groups. The control group will undergo a simulation training session without music, while the intervention arm will listen to a Mozart piano sonata during their session. The aim of this study is to determine how listening to Mozart music during surgical simulation training influences learner technical skill acquisition and transfer, as well as their emotions and cognitive load.

DETAILED DESCRIPTION:
Background: The Intelligent Continuous Expertise Monitoring System (ICEMS) is a deep learning application that was developed at the Neurosurgical Simulation and Artificial Intelligence Learning Centre to improve neurosurgical education. The ICEMS assesses and trains bimanual surgical performance by providing continuous feedback via verbal instructions in order to improve trainee performance and mitigate errors. At present, how learners respond to music during surgical training with the ICEMS is unknown.

Rationale: The Mozart effect refers to the short-term enhancement in spatial-temporal reasoning that occurs in learners when they listen to Mozart music. Previous studies have found that exposure to Mozart and/or classical music before or during surgical simulation training can lead to improved performance. However, these studies did not involve a structured artificial intelligence (AI)-enhanced curriculum or objective, quantitative performance assessment based on AI-derived metrics. Moreover, these studies have not assessed how exposure to music during surgical simulation training influences learners' emotions and cognitive load.

This report follows the Consolidated Standards of Reporting Trials-Artificial Intelligence (CONSORT-AI) as well as the Machine Learning to Assess Surgical Expertise (MLASE) checklist.

Hypotheses:

1. Listening to a Mozart piano sonata during surgical simulation training will result in superior skill acquisition and transfer in trainees compared with no music.
2. Listening to a Mozart piano sonata during surgical simulation training will result in lower levels of negative emotions and cognitive load compared with no music.

Primary Objectives: To determine how listening to Mozart music during surgical simulation training influences trainee:

1. Trainee technical skill acquisition and overall surgical performance (composite expertise scores across all practice tasks calculated by the ICEMS).
2. Trainee skill transfer to a more complex realistic scenario (composite expertise scores during realistic task calculated by the ICEMS).

Secondary Objective: To determine how listening to Mozart music during surgical simulation training influences trainee affective-cognitive responses, including emotions-self-reported via questionnaires administered before, during, and after each training session using the Medical Emotions Scale (MES) on 7-point Likert scales-and cognitive load-self-reported via questionnaire administered after each training session using the Cognitive Load Index (CLI) on 5-point Likert scales.

Setting: McGill University's Neurosurgical Simulation and Artificial Intelligence Learning Centre.

Participants: Students enrolled in their preparatory, first, or second year at one of four Quebec medical schools.

Design: A single-blinded two-arm randomized crossover trial.

Intervention: Participants will undergo two separate training sessions of approximately 90 minutes each on the NeuroVR (CAE Healthcare), a virtual reality (VR) surgical simulator that simulates a subpial brain tumor resection. In this study, participants will perform two different scenarios on the NeuroVR: a simple practice scenario and a complex realistic scenario. During each session, participants will perform four repetitions of the practice scenario (5 minutes each) followed by the realistic scenario (13 minutes). The ICEMS will continuously assess performance throughout the trials.

Group 1 (control) will complete their training session without music. Group 2 will listen to Mozart's Sonata for Two Pianos in D Major, K. 448 during their training session.

Verbal feedback will be based on the following six metrics:

1. Tissue injury risk: When a trainee receives feedback on this metric, the healthy brain tissue has been damaged or is at risk of being damaged.
2. Bleeding risk: When a trainee receives feedback on this metric, there is bleeding that must be cauterized or a risk of bleeding.
3. Instrument tip separation distance: Refers to the distance between the tip of the ultrasonic aspirator and the tips of the bipolar forceps. When a trainee receives feedback on this metric, their instruments are too far apart.
4. High bipolar force: Refers to the amount of force applied to the tissue by the bipolar forceps. When a trainee receives feedback on this metric, they are applying too much force with the bipolar.
5. Low bipolar force: Refers to the amount of force applied to the tissue by the bipolar forceps. When a trainee receives feedback on this metric, they are not applying enough force with the bipolar.
6. High aspirator force: Refers to the amount of force applied to the tissue by the ultrasonic aspirator. When a trainee receives feedback on this metric, they are applying too much force with the aspirator.

These metrics will continuously be evaluated by the ICEMS. The ICEMS will only provide feedback on one metric at a time according to a predetermined hierarchy (in the order listed above). For example, if the ICEMS detects on error on both bleeding risk (2) and high aspirator force (6) at the same time, the system will only provide feedback on bleeding risk since this metric is above high aspirator force in the hierarchy.

Study Procedure: Prior to the simulation session, the study coordinator will stratify participants according to their year in medical school and block randomize them to one of three intervention arms with an allocation ratio of 1:1. Upon arrival, participants will read and sign an informed consent form. They will then fill out a pre-trial questionnaire recording demographic information and self-reported baseline emotions using the MES. Trial instructions introducing the NeuroVR simulator, the instruments, and the practice subpial resection scenario will be provided via a written document. Each practice task will last 5 minutes, followed by a 5-minute rest period. No post-hoc feedback will be provided during the rest periods. Participants will perform their first practice task without feedback to establish a baseline. Participants will then perform their second through fourth practice tasks while receiving metric-specific verbal feedback from the ICEMS. During these formative practice tasks, music will be turned on for the experimental group and paused during the rest periods. Following the completion of the practice tasks, participants will complete a peri-trial questionnaire to assess their emotions using the MES. They will be provided with another information document introducing the realistic subpial brain tumor resection task. Participants will complete the 13-minute realistic task to assess their skill transfer to a more complex scenario. Finally, they will fill out a post-trial questionnaire assessing their emotions using the MES and their cognitive load using the CLI.

ELIGIBILITY:
Inclusion Criteria:

* Medical students who are actively enrolled in their preparatory, first, second year of medical school at any Quebec institution who do not fit the exclusion criteria.

Exclusion Criteria:

* Prior use of the NeuroVR (CAE Healthcare) simulator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Intelligent Continuous Expertise Monitoring System (ICEMS) expertise score - Technical skill acquisition across practice tasks on NeuroVR simulator | 1 day of study
  The ICEMS will continuously evaluate the trainee's performance during each practice task and calculate average expertise scores on a scale of -1.00 (novice) to 1.00 (expert). This will allow us to assess learner technical skill acquisition from the first through fifth repetitions of the practice task.
Intelligent Continuous Expertise Monitoring System (ICEMS) expertise score - Technical skill transfer during complex realistic task on NeuroVR simulator | 1 day of study
  The ICEMS will continuously evaluate the trainee's performance during the realistic task and calculate an average expertise score on a scale of -1.00 (novice) to 1.00 (expert). This will allow us to assess learner technical skill transfer from the practice tasks to a more complex realistic scenario.

SECONDARY OUTCOMES:
Strength of emotions elicited | 1 day of study
  Measured using Duffy's Medical Emotions Scale (MES) before, during, and after learning (self-reported via questionnaires on 7-point Likert scales).
Levels of cognitive load | 1 day of study
  Measured using Leppink's Cognitive Load Index (CLI) after learning (self-reported via questionnaire on 5-point Likert scales).

CONTACTS AND LOCATIONS:
Overall Officials: Rolando F. Del Maestro, MD, PhD, Principal Investigator — Neurosurgical Simulation and Artificial Intelligence Learning Centre
Locations (1):
- Neurosurgical Simulation and Artificial Intelligence Learning Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data obtained from primary and secondary outcomes may be shared if other researchers have an interest in this data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available for 5 years following the completion of the trial.
Access Criteria: Researchers who wish to access the data must contact the principal investigator of the trial, Dr. Rolando F. Del Maestro.

REFERENCES:
- [Background] Duffy MC, Lajoie SP, Pekrun R, Lachapelle K. Emotions in medical education: Examining the validity of the Medical Emotion Scale (MES) across authentic medical learning environments. Learn Instr. 2020;70:101150. doi:10.1016/j.learninstruc.2018.07.001
- [Background] R Core Team. R: A Language and Environment for Statistical Computing. Vienna, Austria: R Foundation for Statistical Computing; 2025. https://www.R-project.org/
- [Background] Leppink J, Paas F, Van der Vleuten CP, Van Gog T, Van Merrienboer JJ. Development of an instrument for measuring different types of cognitive load. Behav Res Methods. 2013 Dec;45(4):1058-72. doi: 10.3758/s13428-013-0334-1. PMID 23572251
- [Background] Winkler-Schwartz A, Bissonnette V, Mirchi N, Ponnudurai N, Yilmaz R, Ledwos N, Siyar S, Azarnoush H, Karlik B, Del Maestro RF. Artificial Intelligence in Medical Education: Best Practices Using Machine Learning to Assess Surgical Expertise in Virtual Reality Simulation. J Surg Educ. 2019 Nov-Dec;76(6):1681-1690. doi: 10.1016/j.jsurg.2019.05.015. Epub 2019 Jun 13. PMID 31202633
- [Background] Liu X, Cruz Rivera S, Moher D, Calvert MJ, Denniston AK; SPIRIT-AI and CONSORT-AI Working Group. Reporting guidelines for clinical trial reports for interventions involving artificial intelligence: the CONSORT-AI extension. Lancet Digit Health. 2020 Oct;2(10):e537-e548. doi: 10.1016/S2589-7500(20)30218-1. Epub 2020 Sep 9. PMID 33328048
- [Background] Wiseman MC. The Mozart effect on task performance in a laparoscopic surgical simulator. Surg Innov. 2013 Oct;20(5):444-53. doi: 10.1177/1553350612462482. Epub 2012 Nov 14. PMID 23154636
- [Background] Nees LK, Grozinger P, Orthmann N, Rippinger N, Hennigs A, Sohn C, Domschke C, Wallwiener M, Rom J, Riedel F. The Influence of Different Genres of Music on the Performance of Medical Students on Standardized Laparoscopic Exercises. J Surg Educ. 2021 Sep-Oct;78(5):1709-1716. doi: 10.1016/j.jsurg.2021.03.008. Epub 2021 Mar 31. PMID 33812805
- [Background] Rauscher FH, Shaw GL, Ky KN. Listening to Mozart enhances spatial-temporal reasoning: towards a neurophysiological basis. Neurosci Lett. 1995 Feb 6;185(1):44-7. doi: 10.1016/0304-3940(94)11221-4. PMID 7731551
- [Background] Yilmaz R, Winkler-Schwartz A, Mirchi N, Reich A, Christie S, Tran DH, Ledwos N, Fazlollahi AM, Santaguida C, Sabbagh AJ, Bajunaid K, Del Maestro R. Continuous monitoring of surgical bimanual expertise using deep neural networks in virtual reality simulation. NPJ Digit Med. 2022 Apr 26;5(1):54. doi: 10.1038/s41746-022-00596-8. PMID 35473961